CLINICAL TRIAL: NCT03035643
Title: Dissected Aorta Repair Through Stent Implantation (DARTS): A Feasibility Study
Brief Title: DARTS I Feasibility Study
Acronym: DARTS I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascyrus Medical LLC. (Industry)
Collaborators: Artivion Inc. (Industry)
Responsible Party: Sponsor
Organization: Artivion Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00066039_AME3
Record Dates: First submitted 2017-01-20; First posted 2017-01-30 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Aortic Dissection; Intramural Hematoma
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, non-blinded, single-arm study evaluating the feasibility and safety of AMDS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMDS Implantation (Experimental): AMDS implantation is performed during an open chest procedure for intervention of aortic dissection repair.
  Interventions: Device: AMDS

INTERVENTIONS:
Device: AMDS — The device will be implanted during an already planned surgical intervention for aortic dissection repair. The participant will be observed and data gathered during the surgery and routine standard of care follow up visits.

SUMMARY:
The objective of this study is to investigate the feasibility and clinical benefits of the AMDS to treat patients with acute DeBakey type I dissections and/or intramural hematomas (IMH) involving the ascending aorta and aortic arch through open surgical repair.

DETAILED DESCRIPTION:
AMDS is designed to complement the replacement of the ascending aorta with conventional surgical technique utilizing a conventional polyester graft. AMDS is constructed of an uncovered Nitinol wire braided stent attached proximally to a polytetrafluoroethylene (PTFE) felt graft component. The PFTE felt graft component excludes the FL at the distal aortic anastomosis and the wire stent re-expands the dissection flap within the arch and descending aorta, which aims to treat malperfusion and promote positive remodeling of the aorta.

The DARTS I Feasibility study is a prospective, non-randomized, non-blinded, single-arm, multi-institutional Canadian study evaluating the feasibility and safety of the AMDS graft. A goal of 40 subjects will be enrolled at approximately 5 sites in Canada.

The enrollment period will span a minimum of 12 months from Institutional Review Board (IRB) approval and site activation. Candidates for this study are adults who require repair of an acute DeBakey type I aorta dissection and/or intramural hematoma (IMH). Patients will be consented pre-operatively and enrolled patients will be followed for approximately 5 years after their AMDS implantation date. Data will be collected at 10 time points: baseline (pre-operatively), discharge, 1 month post-operatively, 3 months post-operatively, and 6 months post-operatively, 1 year post-operatively and thereafter, annually, for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

Subject must have one of the following diagnosed, based on CT angiography, within 0-14 days:

1. Acute DeBakey type I dissection or
2. Acute DeBakey type I intramural hematoma (IMH)

Exclusion Criteria:

General Exclusion Criteria

Patients must be excluded from the study if any of the following conditions are true:

1. Less than 18 years of age or over 80 years of age
2. Life expectancy less than 2 years
3. Pregnant or breastfeeding or planning on becoming pregnant within 60 months
4. Unwilling to comply with the follow-up schedule
5. Refusal to give informed consent

Medical Exclusion Criteria

Patients must be excluded from the study if any of the following conditions are true:

1. Uncontrolled systemic infection
2. Uncontrollable anaphylaxis to iodinated contrast
3. Known allergy(ies) to Nitinol and/or PTFE
4. Patient in extreme hemodynamic compromise requiring cardiopulmonary resuscitation (CPR)
5. Inability to obtain CT angiograms for follow-up
6. Previously diagnosed with Marfan syndrome, Loeys- Dietz syndrome or Ehlers- Danlos syndrome with confirmed laboratory genetic testing on a date prior to the diagnosis of the dissection

Anatomical Exclusion Criteria

1. Any pathology of mycotic origin
2. Subacute or chronic dissection of the ascending aorta and aortic arch (>14 days after the index event)
3. Aortic fistulous communication with non-vascular structure (e.g. esophagus, bronchial)
4. Extensive thrombus or calcifications in the aortic arch as defined by CT angiography
5. Excessive tortuosity precluding safe passage of the AMDS as defined by CT angiography
6. Descending thoracic aneurysm involving the proximal third (1/3) of the descending aorta and measuring > 45mm in diameter.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with device-related mortality | Early (within 30 days)
  The number of patients with mortality related to the treatment device
Number of participants with device-related mortality | Intermediate (3 months)
  The number of patients with mortality related to the treatment device
Number of participants with device-related mortality | Late (6 months)
  The number of patients with mortality related to the treatment device
Number of participants with neurological complications (TIA, stroke) | Early (within 30 days)
  The number of patients with neurological complications related to the treatment device
Number of participants with neurological complications (TIA, stroke) | Intermediate (3 months)
  The number of patients with neurological complications related to the treatment device
Number of participants with neurological complications (TIA, stroke) | Late (6 months)
  The number of patients with neurological complications related to the treatment device

SECONDARY OUTCOMES:
Thrombosis of the false lumen within the confines of the device | Annually, through study completion, an average of 5 years
  Efficacy outcome: Number of participants with false lumen exclusion within the treatment area confined by the treatment device.
Assess need for stent removal | Annually, through study completion, an average of 5 years
  Stent placement and retention. The number of patients requiring removal of the stent.
Successful reattachment of the intimal flap within the arch | Annually, through study completion, an average of 5 years
  The number of patients that has successful reattachment of the intimal flap within the arch following the implantation of AMDS
Successful device deployment, and radiographic evidence of false lumen exclusion within the confines of the device | Annually, through study completion, an average of 5 years
  The number of patients which has successful AMDS deployment and which also had radiographic evidence of false lumen exclusion within the confines of AMDS

OTHER OUTCOMES:
Aortic injury associated with the implantation of the device | Annually, through study completion, an average of 5 years
  The number of patients which has any aortic injury(ies) associated with the implantation of AMDS
Aortic arch branch vessel patency | Annually, through study completion, an average of 5 years
  An evaluation of the patency of aortic arch branch vessels for patients which have had AMDS implantation. Aortic arch branch vessel patency will be evaluated by CTA with a Core Imaging Lab.
AMDS related re-interventions after the dissection repair | Annually, through study completion, an average of 5 years
  The number of patients which have required re-interventions related to the AMDS implantation following the index procedure for aortic dissection repair.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Forcillo, MD, Principal Investigator — Centre Hospitalier de I'Universite de Montreal; Maral Ouzounian, MD, Principal Investigator — University Health Network - Toronto General Hospital; Michael Chu, MD, Principal Investigator — London Health Science Center; Philippe Demers, Principal Investigator — Montreal Heart Institute; Michael Moon, MD, Principal Investigator — University of Alberta
Locations (5):
- Canada (5):
  - Mazankowski Alberta Heart Institute, University of Alberta, Edmonton, Alberta
  - London Health Sciences Center- University Hospital, London, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de I'Universite de Montreal (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozso SJ, Nagendran J, Chu MWA, Kiaii B, El-Hamamsy I, Ouzounian M, Kempfert J, Starck C, Moon MC. Midterm Outcomes of the Dissected Aorta Repair Through Stent Implantation Trial. Ann Thorac Surg. 2021 Feb;111(2):463-470. doi: 10.1016/j.athoracsur.2020.05.090. Epub 2020 Jul 13. PMID 32673661
- [Background] Bozso SJ, Nagendran J, MacArthur RGG, Chu MWA, Kiaii B, El-Hamamsy I, Cartier R, Shahriari A, Moon MC. Dissected Aorta Repair Through Stent Implantation trial: Canadian results. J Thorac Cardiovasc Surg. 2019 May;157(5):1763-1771. doi: 10.1016/j.jtcvs.2018.09.120. Epub 2018 Oct 26. PMID 30501947
- [Background] Bozso SJ, Nagendran J, Chu MWA, Kiaii B, El-Hamamsy I, Ouzounian M, Kempfert J, Starck C, Shahriari A, Moon MC. Single-Stage Management of Dynamic Malperfusion Using a Novel Arch Remodeling Hybrid Graft. Ann Thorac Surg. 2019 Dec;108(6):1768-1775. doi: 10.1016/j.athoracsur.2019.04.121. Epub 2019 Jun 27. PMID 31254509
- [Background] Montagner M, Kofler M, Heck R, Buz S, Starck C, Kurz S, Falk V, Kempfert J. Initial experience with the new type A arch dissection stent: restoration of supra-aortic vessel perfusion. Interact Cardiovasc Thorac Surg. 2021 Jul 26;33(2):276-283. doi: 10.1093/icvts/ivab085. PMID 34010408